CLINICAL TRIAL: NCT02298907
Title: Cardiopulmonary Exercise Variables Are Associated With Postoperative Morbidity After Major Colorectal Surgery - A Validation Study
Brief Title: CPET in Colorectal Surgery
Status: Completed | Type: Observational
Sponsor: Liverpool University Hospitals NHS Foundation Trust (Other Government)
Collaborators: Medway NHS Foundation Trust (Other); Maidstone & Tunbridge Wells NHS Trust (Other); Torbay and South Devon NHS Foundation Trust (Other); University Hospital Plymouth NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 14/EM/1038
Record Dates: First submitted 2014-06-30; First posted 2014-11-24 (Estimated); Last update posted 2022-06-09 (Actual); Status verified 2015-06

CONDITIONS: Colorectal Cancer; Surgery
Keywords: colorectal cancer; surgery; cardiopulmonary exercise testing; perioperative; fitness
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The present study is a retrospective analysis of prospectively collected clinical data. Anonymized data from patients collected during routine clinical care from 7 major colorectal units in the UK who perform pre-operative cardiopulmonary exercise testing will be pooled at a central location (Aintree University Hospitals, Liverpool) and used to validate the relationship between cardiopulmonary exercise testing (CPET) variables and short term post-operative outcomes after major colorectal surgery. Here the investigators will attempt to validate a study entitled "Cardiopulmonary exercise variables are associated with postoperative morbidity after major colonic surgery - a prospective blinded observational study" previously published by our team in Liverpool .

DETAILED DESCRIPTION:
Patients in all the centres (Aintree University Hospitals NHS Foundation Trust, University Hospital Crosshouse NHS Foundation Trust, Barts Healthcare NHS Foundation Trust, East Kent Hospitals University NHS Foundation Trust, Lancashire Teaching Hospitals NHS Foundation Trust, South Devon Healthcare NHS Foundation Trust and Maidstone and Tunbridge Wells NHS Trust) will undergo a maximal CPET prior to major colorectal surgery (defined as a procedure involving bowel resection +/- an anastomosis or stoma) according to the CPET protocol defined in Appendix 1. If the CPET deviates from this protocol, the centre would need to clear their local CPET protocol with the Principle Investigator (PI). All variables measured by CPET which will be collected are outlined in Appendix 2.

Following the CPET, patients will undergo a major colorectal surgical procedure. Following surgery only routine clinically relevant observational data will be collected. These data will relate to hospital length of stay, the level of care required following surgery, post-operative morbidity (Postoperative Morbidity Survey - POMS and Clavine Dindo Score) and the recovery process. Most of this information can be accessed from prospectively maintained enhanced recovery databases, however patient notes and electronic patient records are acceptable alternatives. Appendix 2 shows the minimum dataset that will be collected.

All data from each individual hospital will be anonymized at source and the PI will only be sent CPET variables, post-operative outcome data, and basic patient demographics (outlined in Appendix 2) which cannot be linked back to the original patient.

We aim to include all patients aged >18 years considered for major colorectal surgery (benign or malignant) and undergoing an enhanced recovery programme after surgery. Patients will be excluded if they have diagnosis of inflammatory bowel disease, patients scheduled for neoadjuvant cancer therapy, patients physically unable to perform a CPET on a cycle ergometer, patients having no surgery performed or interim emergency surgery, patients lacking complete in-hospital morbidity data. All patients received an information sheet regarding CPET and written consent for the CPET as part of their routine care was obtained at each centre.

Hypothesis

This study tests the hypothesis that CPET variables are related to short-term in-hospital morbidity in patients undergoing major colorectal surgery.

Our primary aim is to establish a reliable relationship between post-operative complications (present or absent) and oxygen uptake (Vo2) at estimated lactate threshold (LT); a secondary aim is to explore the multivariable relationship between CPET variables and other important prognostic variables with post-operative complications in an attempt to risk stratify patients before major surgery.

Statistical methods

Non-parametric receiver operator characteristic (ROC) curves were constructed for Vo2 at LT, Vo2 at Peak, O2 Pulse at LT and ventilatory equivalents for carbon dioxide (VE/ co2 at LT) in order to assess their independent ability to discriminate between patients with and without post-operative morbidity. Optimal cut-points will be obtained by minimising the distance between points on the ROC curve and the upper left corner. Six variables (to satisfy the 10 events per variable rule (26)) were identified as candidates for a multivariable logistic regression model: Vo2 at LT and at Peak, gender, operation type (laparoscopic/open), and O2 Pulse at LT and VE/ co2 at LT. A final multivariable model will be obtained using forward stepwise selection (minimising Akaike Information Criteria (AIC)). Its sensitivity to variable exclusion and re-inclusion will also be assessed using AIC. Model fit will be assessed using the Hosmer-Lemeshow goodness-of-fit test. In order to explore the univariate relationship between CPET variables and length of stay, continuous CPET variables will be dichotomised at the optimal cut-point for the ROC curve and Kaplan-Meier curves will be constructed. The log rank test will be used to compare survival curves; patients who died before discharge will be treated as right-censored. Patients who are discharged before day 5 will be excluded from the analysis of length of stay. All analyses will be conducted using Stata (StataCorp. 2011 Stata Statistical Software: Release 12. College Station, TX: StataCorp LP.). Continuous variables will be reported as mean and standard deviation (SD) or median and inter-quartile range (IQR) depending on the distribution. Categorical variables will be presented as frequency (percentage). P-values will be obtained using univariate logistic regression (continuous) and Chi-squared or Fisher's Exact tests (categorical). Statistical significance will be taken at 5%.

We aim to recruit 500 patients who will undergo a CPET, elective colorectal surgery and post-operative follow-up. For a hypothesised AUROC of 0.63, based on our previous study, 500 patients would be required to demonstrate that Vo2 at LT is better than chance at discriminating between patients with and without post-operative morbidity. This estimate is based on a 5-day morbidity incidence of 48%, 90% power and a two-tailed 5% significance level. The calculated sample size is based on that needed to evaluate the area under the ROC curve (AUROC).

Appendix 1

Pulmonary Function Tests (PFT's)

The patients will perform pulmonary function tests (breathing tests). The breathing tests will be performed before the CPET.

Cardiopulmonary Exercise Testing

A symptom limited CPET will be performed as part of patients routine care occurring before surgery. Specifically, this involves cycling on an exercise bike for 8-12 minutes. Starting with a very low resistance on the pedals the patient will pedal at 60 revolutions per minute. After 3 minutes of cycling, the resistance will gradually increase at a constant rate until the patient can no longer turn the pedals at the required speed. The patient's heart will be monitored by an electrocardiogram (ECG). The patient will wear a soft rubber mask in order to continuously sample expired air with an online breath by breath gas analyser. This test is common practice prior to operations and provides an accurate measure of physical capacity and each centre involved in data pooling have similar CPET protocols as described above. Each CPET appointment lasts approximately one hour, however this is always part of routine car. BORG scores will be assessed at intervals as per local policy.

CPET will follow American Thoracic Society/ American College of Chest Physicians recommendations (27). Ventilation and gas exchange variables are measured using a metabolic cart. Pulse, 12-lead ECG, blood pressure and pulse oximetry will be monitored throughout. Ramp gradient will be set to 10-25 W/min based on a calculation (28) using predicted freewheel oxygen uptake ( o2), predicted o2 at peak exercise, height and age. Any major adverse clinical events occurring during CPET will be documented.

Measurements

Patient characteristics are recorded as per Appendix 2. Resting flow-volume loops will be used to derive Forced Expiratory Volume over 1 second (FEV1) and Forced Vital Capacity (FVC). Ventilation and gas exchange variables derived from CPET included Vo2, ventilatory equivalents for oxygen and carbon dioxide (VE/ o2; VE/ co2) and oxygen pulse ( o2/heart rate), all measured at LT and at peak exercise (28).

LT will be estimated conventionally (breakpoint in the co2- o2 relationship (29), with increases in VE/ o2 and end tidal (PET) O2 but no increase in VE/ co2 or decrease in PET co2 (30). Peak Vo2 will be averaged over the last 30 seconds of exercise. CPETs will be reported by an experienced assessor usually an experiences exercise physiologist or consultant anaesthetist.

Appendix 2

Short-term surgical outcome will assessed as morbidity (by medical and nursing staff blind to any CPET data) using the 9 domains listed in the Post-Operative Morbidity Survey (31) on day 3,5,7 and 14 as well as the Clavien-Dindo Classification (32) (highest grade for the most serious sustained in-hospital complication) and in-hospital mortality.

Length of hospital stay (days) will be recorded. All patients are usually followed for 30 days post-discharge for re-admission and mortality however this is not essential.

All information collected following surgery will be carried out by observation only.

List of Measurements that will be collected during tests and post-operative follow-up

List of derived variables from CPET and Spirometry

Baseline demographics

* Age
* Gender
* Height
* Weight
* Diagnosis
* Planned operation type
* Pre-existing diagnosis of diabetes, ischaemic heart disease, cerebrovascular disease, or heart failure.
* Staging (if malignancy
* WHO classification
* American Society of Anesthesiologists - Physical Status Scores (ASA-PS)

Prior to test, Spirometry for:

* Forced Expiratory Volume in 1 Second (FEV1)
* Forced Vital Capacity (FVC)
* Calculated MVV (FEV1 * 40).

Cardio-respiratory and work variables recorded at rest and continuously throughout the test:

* Heart rate (HR)
* Blood pressure (BP)
* Oxygen saturation (SaO2)
* Tidal volume (Vt)
* Respiratory rate (RR)
* Minute ventilation (Vt*RR)
* Work rate (in Watts, from cycle ergometer)

Measures of Exercise capacity

* Lactate threshold (LT): absolute and ml/Kg
* Peak Oxygen consumption (VO2 peak): absolute and ml/Kg

Indicators suggestive of cardiac limitation to exercise capacity at LT:

* Oxygen pulse at LT
* Early ischaemia (before LT) on 12-lead ECG

Indicators suggestive of cardiac limitation to exercise capacity at Vo2 peak:

* HR reserve at Vo2 peak
* Late ischaemia (after LT) on 12-lead ECG

Ventilatory equivalent for VO2 ( VE/ o2) and CO2 ( VE/ co2)

* at LT
* at Vo2 Peak
* Calculated using the slope of the relationship throughout the CPET test

Oxygen pulse at LT and Vo2 Peak

AND:

Vo2/WR slope

List of post-operative outcome data

Post-Operative Morbidity Survey (POMS) collected at day 3, 5, 7 and 14 post-surgery

Clavien-Dindo score Hospital Resource utilization - Length of hospital stay (days) If available - 30-day mortality, 30-day readmission rate

ELIGIBILITY:
Inclusion Criteria:

* all patients aged >18 years considered for major colorectal surgery (benign or malignant) and undergoing an enhanced recovery programme after surgery

Exclusion Criteria:

* patients scheduled for neoadjuvant cancer therapy, patients physically unable to perform a CPET on a cycle ergometer, patients having no surgery performed or interim emergency surgery, patients lacking complete in-hospital morbidity data.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive colorectal cancer patients recruited via colorectal multidisciplinary meeting
Sampling Method: Non-Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2010-06; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Oxygen uptake at lactate threshold | baseline

SECONDARY OUTCOMES:
Oxygen uptake at peak | baseline
Power output at lactate threshold and peak exercise | baseline
Ventilatory equivalents at lactate threshold and peak exercise | baseline
Number of patients with adverse post-operative outcome measures | post-operatively

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm West, Principal Investigator — Aintree University Hospitals NHS
Locations (1):
- Aintree University Hospital, Liverpool, United Kingdom

REFERENCES:
- [Background] West MA, Lythgoe D, Barben CP, Noble L, Kemp GJ, Jack S, Grocott MP. Cardiopulmonary exercise variables are associated with postoperative morbidity after major colonic surgery: a prospective blinded observational study. Br J Anaesth. 2014 Apr;112(4):665-71. doi: 10.1093/bja/aet408. Epub 2013 Dec 8. PMID 24322573